CLINICAL TRIAL: NCT00321750
Title: Phase 2 Study of the Treatment of Oral Erosive Lichen Planus With 1% Pimecrolimus Cream: a Double Blind Randomized Prospective Trial With Measurement of Pimecrolimus Levels in the Blood
Brief Title: Treatment of Oral Erosive Lichen Planus With Pimecrolimus Cream
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CFR01
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-05

CONDITIONS: Oral Erosive Lichen Planus
Keywords: Oral erosive lichen planus; pimecrolimus cream
MeSH Terms: interventions — pimecrolimus

INTERVENTIONS:
Drug: 1% pimecrolimus cream

SUMMARY:
Background and hypothesis. Oral erosive lichen planus (OELP) is a severe form of mucosal lichen planus. Lesions often induce intense pain and limit feeding. Its course is chronic with flares and spontaneous remissions are rare. Treatment is difficult: topical steroids are usually used first but antimalarials, oral retinoids, systemic steroids, immunosuppressive drugs and even extracorporeal photochemotherapy can be necessary for treating severe forms. The need for novel therapies with less morbidity is obvious. Calcineurin inhibitors have a theoretical interest in treating OELP: this has been emphasized by several open studies performed with topical tacrolimus. The effectiveness of 1% pimecrolimus cream has been suggested by a few case reports and by one recent comparative study which confirmed the potential interest of topical pimecrolimus in treating OELP. The absorption of pimecrolimus through human mucosa is still unknown. Its application on ulcerative lesions such as OELP ones, could lead to significant systemic levels of the molecule.

Objective: To evaluate the efficacy of 1% pimecrolimus cream in treating oral erosive lichen planus (OELP) and to assess its tolerance.

DETAILED DESCRIPTION:
Background and hypothesis. Oral erosive lichen planus (OELP) is a severe form of mucosal lichen planus. Lesions often induce intense pain and limit feeding. Its course is chronic with flares and spontaneous remissions are rare. Treatment is difficult: topical steroids are usually used first but antimalarials, oral retinoids, systemic steroids, immunosuppressive drugs and even extracorporeal photochemotherapy can be necessary for treating severe forms. The need for novel therapies with less morbidity is obvious. Calcineurin inhibitors have a theoretical interest in treating OELP: this has been emphasized by several open studies performed with topical tacrolimus. The effectiveness of 1% pimecrolimus cream has been suggested by a few case reports and by one recent comparative study which confirmed the potential interest of topical pimecrolimus in treating OELP. The absorption of pimecrolimus through human mucosa is still unknown. Its application on ulcerative lesions such as OELP ones, could lead to significant systemic levels of the molecule.

Objective: To evaluate the efficacy of 1% pimecrolimus cream in treating oral erosive lichen planus (OELP) and to assess its tolerance.

Design: Double blind randomized trial with placebo control.

Settings: Outpatients of the Department of Dermatology of the University hospital of Nice, France.

Patients: Fourteen consecutive patients with OELP confirmed by histological examination and with a clinical score superior to 3. 1% pimecrolimus cream or its vehicle were applied on ulcerated lesions twice a day for 4 weeks.

Main outcome measures; the efficacy of the treatment was quantified using a 12 points clinical score. Blood level of pimecrolimus was analyzed at D0, D14 and D28.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the diagnosis of OELP by histological examination and a clinical score superior to 3

Exclusion Criteria:

* Patients under 18 years
* Pregnancy or breast feeding
* Malignancy
* Severe or recurrent infections
* Uncontrolled chronic disorders
* Congenital or acquired immunosuppression and concomitant treatments potentially effective on OELP such as antimalarials, oral retinoids, steroids or immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 2004-12; Study Completion 2005-04

PRIMARY OUTCOMES:
The efficacy of the treatment was quantified using a 12 points clinical score.
Blood level of pimecrolimus was analyzed at D0, D14 and D28.

SECONDARY OUTCOMES:
Side effects
Complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: Thierry D Passeron, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice; Jean-Philippe Lacour, MD, Study Director — Centre Hospitalier Universitaire de Nice; Jean-Paul Ortonne, MD, Study Chair — Centre Hospitalier Universitaire de Nice; Eric Fontas, MD, Study Chair — Centre Hospitalier Universitaire de Nice

REFERENCES:
- [Derived] Passeron T, Lacour JP, Fontas E, Ortonne JP. Treatment of oral erosive lichen planus with 1% pimecrolimus cream: a double-blind, randomized, prospective trial with measurement of pimecrolimus levels in the blood. Arch Dermatol. 2007 Apr;143(4):472-6. doi: 10.1001/archderm.143.4.472. PMID 17438179